CLINICAL TRIAL: NCT07255755
Title: A Double Blind Randomised Clinical Study to Evaluate Attention Improvement in an Adult Population After Cereboost Intake
Brief Title: Cereboost (American Ginseng Extract) and Brain Function
Acronym: REACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Givaudan France Naturals (Industry); Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: R211952; IRAS355890 (Other: Health Research Authority (HRA))
Record Dates: First submitted 2025-11-14; First posted 2025-12-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Attention; Cognition
Keywords: American Ginseng; Cereboost
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): A placebo capsule (containing maltodextrin)
  Interventions: Dietary Supplement: Placebo product
- Study Product (Experimental): Study product capsule containing 200mg American Ginseng extract (Cereboost TM)
  Interventions: Dietary Supplement: American Ginseng extract

INTERVENTIONS:
Dietary Supplement: American Ginseng extract — Cereboost TM capsules delivering 200 mg of Panax quinquefolius extract standardised for ginsenosides (10-12%)
  Arms: Study Product
Dietary Supplement: Placebo product — Placebo capsules, identical in appearance to active treatment, but only containing maltodextrin
  Arms: Placebo

SUMMARY:
The study will assess the immediate, short-term benefits of a single dose of a supplement containing 200mg of Panax quinquefolius (American Ginseng) on cognition (brain function) in healthy young adults.

To understand the effect this product may have, the participants will complete a series of questionnaires and cognitive tests (tests of memory and brain function) at set intervals across a 6-hour period. Blood samples will also be collected to assess the impact of the study product on the participants.

DETAILED DESCRIPTION:
Lifestyle strategies such as nutritional interventions have received increased attention as they provide safe and effective solutions to improve cognitive performance. Ginseng, a popular herbal root extract obtained from plants of the Panax family, is widely regarded as a panacea in traditional medicine and has been used for centuries to treat mental and physical ailments and promote longevity. Ginseng contains a number of bioactives including flavonoids and other phenolic compounds, essential oils, and vitamins. However, the main bioactive ingredients in ginseng are purported to be ginsenosides including Rb1, Re, Rd, and F11. Among multiple species of ginseng, American ginseng (Panax quinquefolius) provides a particularly rich source of these ginsenoside when compared to other ginseng varieties, and emerging research suggests that supplementation with Panax quinquefolius may elicit cognitive enhancement effects.

Cereboost TM from Givaudan SA is a standardised extract of American ginseng and has been reported to exert such benefits. For example, following acute supplementation with 100 mg, 200 mg and 400 mg Cereboost TM, improvements on an immediate word recall task, a visuospatial working memory task, a choice reaction time task, a composite working memory factor, and a measure of subjective mood (i.e. calmness) were observed in healthy young adults (aged 18-40 years) during the six hours after consumption. Adding to these findings, a study of middle-aged adults (aged 40-60 years) observed similar acute benefits of 200 mg Cereboost TM on a composite working memory factor after three hours, although no changes in mood were observed in this older age group. More recently, improved working memory and attention during the immediate postprandial period (2-6 hours) in healthy young adults was reported following Cereboost TM 200mg intake.

We are interested in conducting a larger study (n=200) employing standardised methods to investigate the acute benefits of a single dose (200mg) of American ginseng (Cereboost TM) and focusing mainly on the Modified Attention Network Task (MANT) test as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, the Participant must fulfil all the following criteria:

1. Be able to give written informed consent.
2. Be between 18-40 years, inclusive.
3. Depression Anxiety and Stress Scale scores (DASS-21):

   1. Depression ≤9
   2. Anxiety ≤7
   3. Stress ≤14
4. Willing to refrain from alcohol consumption 24-hours prior to assessment visits.
5. Willing to refrain from caffeine consumption (including but not limited to energy drinks, soda, coffee…) on the morning of the assessment visit.
6. Non-smokers and non-vapers
7. Willing to consume the Study Product (SP).
8. Willing to attend the study visit in an overnight fasted state, having followed a low-polyphenol diet for 48 h.
9. Fluent in written and spoken English

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

1. Participants who are pregnant or wish to become pregnant during the study or who are lactating and/or currently breastfeeding.
2. Has food allergies or other issues with foods that would preclude intake of the Study Products.
3. Not willing to consume gelatine from bovine/porcine source
4. Has a BMI ≤18.5 or ≥30kg/m2
5. Blood pressure >140/90 mmHg
6. Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results.
7. Excluded health conditions include:

   1. Cognitive disorders in the past 12 months.
   2. Current or past history of a major neuropsychiatric disorder, including: bipolar disorder, schizophrenia and schizotypal personality disorder
   3. Current or past history of a major neurological condition.
   4. Gastrointestinal disorders (e.g. IBS/IBD)
   5. ADHD (attention deficit hyperactivity disorder)
   6. Learning disabilities and difficulties
   7. Current, uncorrected, vision or hearing impairment
8. Current or recent use of a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results. Prohibited medications include:

   1. Anti-psychotics
   2. Anti-coagulants (including Warfarin)
   3. Anti-platelets (including Aspirin and Clopidogrel)
   4. Sedatives
   5. Monoamine Oxidase Inhibitors (MAOIs)
9. Taking any dietary supplements and unwilling to stop for two weeks prior to and for the duration of participation in the study
10. Current or history of drug or alcohol abuse
11. Current or history of: HIV, kidney disease, liver or biliary disorders, cancer, cardiovascular disease, pulmonary disease (chronic respiratory trouble)
12. Planned surgery within 2 weeks of their participation in the study
13. Do not agree to the GP being contacted about participation and screening results
14. Participated in any other cognitive trials within the last month

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Measure of Attention | Baseline, 2-hours, 4-hours and 6-hours post intervention
  Measured by the Attentional Network Task (ANT), expressed by accuracy score (%correct) at 6 hours post consumption

SECONDARY OUTCOMES:
Measure of Cognition (Executive function) | Baseline, 2-hours, 4-hours and 6-hours post intervention
  Measured by a neuropsychological test battery (https://neuropsychology.online) including the following cognitive tasks; Reaction time, Digit span - backwards, Go/No-Go, Spatial working memory - forwards, Trail making B.
Measure of Cognition (Reaction Time) | Baseline, 2-hours, 4-hours and 6-hours post intervention
  Measured by a neuropsychological test battery (https://neuropsychology.online) including the following cognitive tasks; Reaction time, Digit span - backwards, Go/No-Go, Spatial working memory - forwards, Trail making B.
Measure of Mood State | At the beginning and end of the cognitive task batteries at baseline, and at 2-hours, 4-hours and 6-hours post intervention
  Established by the Positive and Negative Affect Schedule - Now (PANAS-X) questionnaire. The questionnaire includes 20 mood-related adjectives, and participants rate the extent to which they are currently experiencing each emotion on a 5-point Likert scale, ranging from 'Very slightly or not at all' (scored as 1) to 'Extremely or very much' (scored as 5).
  Half of the presented words related to positive emotions, the other half to negative emotions. Separate scores are obtained for positive affect and negative affect by summing ratings for all similar emotions.
Measure of Subjective Sleepiness | At the beginning and end of the cognitive task batteries at baseline, and at 2-hours, 4-hours and 6-hours post intervention
  Established by using the validated Karolinska sleepiness scale (KSS), a 9-point Likert scale. Anchor points on the scale are '1. Extremely alert' and '9. Extremely sleepy, it is an effort to stay awake'.
Measure of Subjective Mental Fatigue | At the beginning and end of the cognitive task batteries at baseline, and at 2-hours, 4-hours and 6-hours post intervention
  Established by the subjective mental fatigue questionnaire on a 9-point Likert scale. Anchor points on the scale are '1. Very low/Alert' and '9. Very high/Fatigued'.
Measure of American Ginseng metabolites | Blood collection at 6-hours post intervention timepoint
  Blood sample will be collected to measure metabolites resulting from American ginseng metabolism

CONTACTS AND LOCATIONS:
Overall Officials: David Vauzour, PhD, Principal Investigator — University of East Anglia
Locations (2):
- United Kingdom (2):
  - Quadram Insitute Clinical Research Facility, Norwich, Norfolk
  - University of East Anglia, Norwich, Norfolk

IPD SHARING:
Plan to Share IPD: No